CLINICAL TRIAL: NCT03447821
Title: Efficacy and Safety of CB-01-11 200mg Tablets in Infectious Diarrhoea. A Pilot, Dose Finding, Double-blind, Randomized, Multicentre Study
Brief Title: Efficacy and Safety of CB-01-11 200mg Tablets in Infectious Diarrhoea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cosmo Technologies Ltd (Industry)
Responsible Party: Sponsor
Organization: Cosmo Pharmaceuticals NV (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CB-01-11/03
Record Dates: First submitted 2018-02-09; First posted 2018-02-27 (Actual); Results first posted 2018-10-09 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Infectious Diarrhoea
Keywords: Infectious diarrhoea; rifamycin SV; rifamycin SV MMX; MMX
MeSH Terms: conditions — Dysentery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 400 mg Rifamycin SV dosage (Active Comparator): Two enteric coated, modified release tablets, each containing 200 mg Rifamycin SV, taken three times daily. Four of the six daily tablet taken in this group were placebos.
  Interventions: Drug: 400 mg Rifamycin SV dosage
- 800 mg Rifamycin SV dosage (Active Comparator): Two enteric coated, modified release tablets, each containing 200 mg Rifamycin SV, taken three times daily. Two of the six daily tablet taken in this group were placebos.
  Interventions: Drug: 800 mg Rifamycin SV dosage
- 1200 mg Rifamycin SV dosage (Active Comparator): Two enteric coated, modified release tablets, each containing 200 mg Rifamycin SV, taken three times daily. None of the six daily tablet taken in this group were placebos.
  Interventions: Drug: 1200 mg Rifamycin SV dosage

INTERVENTIONS:
Drug: 400 mg Rifamycin SV dosage
  Arms: 400 mg Rifamycin SV dosage
Drug: 800 mg Rifamycin SV dosage
  Arms: 800 mg Rifamycin SV dosage
Drug: 1200 mg Rifamycin SV dosage
  Arms: 1200 mg Rifamycin SV dosage

SUMMARY:
To assess the safety and the preliminary efficacy data on the three doses of the new Cosmo Technologies oral rifamycin SV colon-release 200 mg tablets manufactured according to MMX technology (CB-01-11) in the treatment of infectious diarrhoea.

DETAILED DESCRIPTION:
To assess the safety and the preliminary efficacy data on the three doses of the new Cosmo Technologies oral rifamycin SV colon-release 200 mg tablets manufactured according to MMXTM technology (CB-01-11) in the treatment of infectious diarrhoea.

Primary end points to determine:

• The safety and preliminary efficacy data of the three doses of the new rifamycin SV formulation tested based upon the time elapsed from the ingestion of the 1st dose of study medication to the passage of the last unformed stool (TLUS), in compliance with the relevant guidelines

Secondary end-points to determine:

* The number of patients showing improvement in diarrhoea during a 24-h interval, i.e. >50 % reduction of bowel movements.
* The number of unformed stools passed per 24-h interval, after dosing.
* The number of patients who are declared to be "well". Wellness is defined as the patient having 48 hours with no unformed stools, a maximum of two soft stools and no clinical symptoms of infectious diarrhoea.
* The number of treatment failures. A treatment failure is defined as clinical deterioration or worsening of symptoms or illness continuing after 120 h following the first dose.
* The number and percentage of patients recovered from diarrhoea. Patients were considered to have recovered if fewer than three unformed stools were passed in the previous 24 hours and no symptom of enteric infection were present.

ELIGIBILITY:
Inclusion Criteria:

Patients had to meet all of the following inclusion criteria:

* Male and female patients aged 18-65 years inclusive on the date of screening.
* Patients with infectious diarrhoea (ID) in the active phase of no more than 72-h duration. Criteria for diagnosis of ID were: three or more unformed stools in the preceding 24 hours, and at least one symptom of enteric infection e.g. abdominal cramps/pain, tenesmus, urgency, an excess of gas/flatulence, nausea, vomiting.
* If female, and of child-bearing potential, use of an effective contraceptive method. (Oral contraceptives, injectable hormonal contraceptives, double-barrier method (condom/diaphragm with spermicide) and intra-uterine devices, according to the definition of Note 3 of ICH M3(M) Guideline. Females were considered not to be of child-bearing potential, if they were at least 12 months post-menopausal.
* Ability, in the investigator's opinion to comprehend the full nature and purpose of the study, including the possible risks and side effects, and willing to comply with the requirements of the study.
* Patients who have voluntarily signed and dated the informed consent document for screening and study specific procedures.
* Patients must be sufficiently literate to be able to complete a diary card.

Exclusion Criteria:

Patients had not to have had of any of the following:

* Females of child-bearing potential not using an effective contraceptive method.
* Pregnant or lactating females.
* Fever (defined as a body (axillary) temperature ≥ 38° C) present either at the screening visit or in the previous 24 hours.
* Visible presence of blood in the stool at baseline.
* Patients with any history or evidence on examination, of clinically significant gastrointestinal (in particular intestinal obstruction and severe intestinal ulcerative lesions), renal, hepatic, endocrine, respiratory, cardiovascular, dermatological or haematological disease, which in the opinion of the investigator could affect the interpretation of the efficacy and safety data.
* Patients with moderate or severe dehydration (see Appendix 2 of the protocol, for definitions of clinical symptoms).
* Prohibited previous and concomitant medication (see relevant section of the protocol).
* History of recent gastrointestinal malignancy (within 6 months).
* Allergy: presumptive or ascertained hypersensitivity to the study drug, history of anaphylaxis or allergic reactions in general.
* History of, or current misuse of alcohol, drugs or abuse of medication.
* Participation in another study with any investigational product within 3 months before screening.
* Patients who, in the opinion of the investigator, could be un-cooperative and/or non-compliant and should not therefore participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Mancera Reyes, Principal Investigator — HOSPITAL CENTRAL DE ORIENTE; Can Polat Eyigün, Principal Investigator — Gülhane Military Medical Academy

IPD SHARING:
Plan to Share IPD: No
None. IPD not to be shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- 400 mg Rifamycin SV Dosage: Two enteric coated, modified release tablets, each containing 200 mg Rifamycin SV, taken three times daily. Four of the six daily tablet taken in this group were placebos.
  400 mg Rifamycin SV dosage
- 800 mg Rifamycin SV Dosage: Two enteric coated, modified release tablets, each containing 200 mg Rifamycin SV, taken three times daily. Two of the six daily tablet taken in this group were placebos.
  800 mg Rifamycin SV dosage
- 1200 mg Rifamycin SV Dosage: Two enteric coated, modified release tablets, each containing 200 mg Rifamycin SV, taken three times daily. None of the six daily tablet taken in this group were placebos.
  1200 mg Rifamycin SV dosage
Period: Overall Study
Arm/Group | 400 mg Rifamycin SV Dosage | 800 mg Rifamycin SV Dosage | 1200 mg Rifamycin SV Dosage
Started | 14 | 13 | 13
Completed | 13 | 12 | 12
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent To Treat
Groups:
- Total: Total of all reporting groups
Arm/Group | 400 mg Rifamycin SV Dosage | 800 mg Rifamycin SV Dosage | 1200 mg Rifamycin SV Dosage | Total
Number analyzed (Participants) | 13 | 12 | 12 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (12.1) | 37.3 (15.9) | 41.9 (12.7) | 39.6 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 7 | 21
  Male | 7 | 4 | 5 | 16
Height (cm) [Mean (Standard Deviation); unit: cm] | 165.2 (9.8) | 160.8 (9.7) | 159.1 (6.2) | 161.8 (8.9)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 72.3 (16.7) | 72.9 (17) | 70.3 (11.8) | 71.8 (15)
Axillary Temperature (°C) [Mean (Standard Deviation); unit: Degrees Celsius] | 36.8 (0.5) | 36.8 (0.4) | 36.7 (0.4) | 36.8 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Time to Last Unformed Stool (TLUS)
Description: The safety and preliminary efficacy data of the three doses of the new rifamycin SV formulation tested based upon the time elapsed from the ingestion of the 1st dose of study medication to the passage of the last unformed stool (TLUS)
Time Frame: Up to 7 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 400 mg Rifamycin SV Dosage | 800 mg Rifamycin SV Dosage | 1200 mg Rifamycin SV Dosage
Number analyzed (Participants) | 13 | 12 | 12
hours | 59.3 (12.1) | 51.4 (12.3) | 57.4 (13.1)

2. Secondary Outcome: The Number of Patients Showing Improvement in Diarrhoea During a 48h Interval
Description: The evaluation of improvement in diarrhoea during a 48 hour interval is defined as a >50% reduction of bowel movements versus the baseline value
Time Frame: 48 hours
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | 400 mg Rifamycin SV Dosage | 800 mg Rifamycin SV Dosage | 1200 mg Rifamycin SV Dosage
Number analyzed (Participants) | 13 | 12 | 12
Participants
  Showed improvement within 48 hrs | 4 | 9 | 6
  Showed no improvement within 48 hrs | 9 | 3 | 6

3. Secondary Outcome: The Number of Unformed Stools Passed Per 24-h Interval
Description: The number of unformed stools passed per 24-h interval, after dosing
Time Frame: 192 hours
Population: ITT
Measure: Mean (Standard Deviation); unit: Unformed stools
Arm/Group | 400 mg Rifamycin SV Dosage | 800 mg Rifamycin SV Dosage | 1200 mg Rifamycin SV Dosage
Number analyzed (Participants) | 13 | 12 | 11
Unformed stools
  0-24 h | 5.23 (2.74) | 4.67 (3.17) | 4.73 (3.41)
  24-48 h | 2.15 (1.95) | 1.5 (1.57) | 2.64 (2.66)
  48-72 h | 2.09 (1.64) | 1.29 (1.6) | 1.7 (1.95)
  72-96 h | 1.5 (1.29) | 1.67 (2.08) | 1.8 (2.05)
  96-120 h | 1.5 (0.71) | 1.5 (2.12) | 0.75 (0.96)
  120-144 h | 3 (0) | 0.5 (0.71) | 1 (0)
  144-168 h | 3 (0) | 1 (0) | 1 (0)
  168-192 h | 0 (0) | 1 (0) | 1 (0)

4. Secondary Outcome: The Number of Patients Who Are Declared to be "Well"
Description: The patient having must meet all of the following criteria in order to be classified as "well": 48 hours with no unformed stools with a maximum of two soft stools and no clinical symptoms of infectious diarrhoea.
Time Frame: 48 hours
Population: intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | 400 mg Rifamycin SV Dosage | 800 mg Rifamycin SV Dosage | 1200 mg Rifamycin SV Dosage
Number analyzed (Participants) | 13 | 12 | 11
Participants
  Wellness Yes | 13 | 10 | 2
  Wellness No | 0 | 2 | 9

5. Secondary Outcome: Number of Participants With Treatment Failure
Description: A treatment failure is defined as clinical deterioration or worsening of symptoms or illness continuing after 120 h following the first dose.
Time Frame: 120 hours
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | 400 mg Rifamycin SV Dosage | 800 mg Rifamycin SV Dosage | 1200 mg Rifamycin SV Dosage
Number analyzed (Participants) | 13 | 12 | 11
Participants
  No | 12 | 10 | 9
  Yes | 1 | 2 | 2

6. Secondary Outcome: The Number of Patients Recovered From Diarrhoea
Description: Patients were considered to have recovered if fewer than three unformed stools were passed in the previous 24 hours and no symptom of enteric infection were present.
Time Frame: 24 hours
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | 400 mg Rifamycin SV Dosage | 800 mg Rifamycin SV Dosage | 1200 mg Rifamycin SV Dosage
Number analyzed (Participants) | 13 | 12 | 11
Participants
  No | 1 | 2 | 2
  Yes | 12 | 10 | 9

ADVERSE EVENTS:
Arm/Group | 400 mg Rifamycin SV Dosage | 800 mg Rifamycin SV Dosage | 1200 mg Rifamycin SV Dosage
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/13 | 3/12 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400 mg Rifamycin SV Dosage (N=13) | 800 mg Rifamycin SV Dosage (N=12) | 1200 mg Rifamycin SV Dosage (N=12)
CARDIAC DISORDERS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Tachycardia
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 2 (2) | 3 (10) | 1 (2)
GENERAL DISORDERS (General disorders) | 2 (2) | 0 (0) | 0 (0)
PSYCHIATRIC DISORDERS (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
SKIN AND SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
NERVOUS SYSTEM (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No disclosure was to take place without written authorisation from Cosmo Technologies Ltd, except to the extent necessary to obtain informed consent from potential volunteers.